CLINICAL TRIAL: NCT05152043
Title: Effects of Romadan Fasting on Variability in Blood Pressure in Healthy and Hypertensive Subjects
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: variability of blood pressure
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
Keywords: Hypertension; Ramadan fasting
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Included participants who have a stable HT who intend to practice RJ

DETAILED DESCRIPTION:
Stable patients with or without diagnosed hypertension that intend to fast ramadan. Each participant is examined during three planned visits. The first takes place during the month preceding Ramadan. The second during the last week of Ramadan and the third thirty days after the end of Ramadan.

Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patients clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with or without diagnosed hypertension intending to fast Ramadan.

Exclusion Criteria :

* Age < 30 years old
* Adult patient with or without diagnosed hypertension not intending to fast Ramadan.

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stable patients with or without diagnosed hypertension that intend to fast ramadan. Each participant is examined during three planned visits. The first takes place during the month preceding Ramadan. The second during the last week of Ramadan and the third thirty days after the end of Ramadan.
  Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patient clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Variability | 60 days
  Values are registered during 24 hours. Diurnal measures are defined as measures conducted during 6 am and 10 pm, whereas nocturnal measures are defined as those registered during the remaining hours. Mean systolic blood pressure and diastolic blood pressure are calculated for the 24 hours for both diurnal and nocturnal period.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia